CLINICAL TRIAL: NCT00714571
Title: Behavioral and Neuroimaging Changes After Cognitive Rehab in TBI and MCI
Brief Title: Behavioral and Neuroimaging Changes After Cognitive Rehab in Traumatic Brain Injuries (TBI) and Mild Cognitive Impairment (MCI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B6366-W
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease; Traumatic Brain Injury
Keywords: cognitive rehabilitation; explicit memory training; mild cognitive impairment; Alzheimer's disease; traumatic brain injury; veterans
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- MST healthy older adults Stage 1 (Active Comparator): Mnemonic strategy training
  Interventions: Behavioral: Mnemonic strategy training (MST)
- MST MCI Stage 1 (Active Comparator): Exposure training
  Interventions: Behavioral: Mnemonic strategy training (MST)
- XP healthy older adults Stage 1 (Active Comparator): XP healthy older adults Stage 1
  Interventions: Behavioral: Repeated exposure (XP)
- XP MCI Stage 1 (Active Comparator): XP MCI Stage 1
  Interventions: Behavioral: Repeated exposure (XP)
- MST healthy older adults Stage 2 (Active Comparator): MST healthy older adults Stage 2
  Interventions: Behavioral: Mnemonic strategy training (MST)
- SCT healthy older adults Stage 2 (Active Comparator): SCT healthy older adults Stage 2
  Interventions: Behavioral: Subtracting Cues training

INTERVENTIONS:
Behavioral: Mnemonic strategy training (MST)
  Arms: MST MCI Stage 1; MST healthy older adults Stage 1; MST healthy older adults Stage 2
Behavioral: Repeated exposure (XP)
  Arms: XP MCI Stage 1; XP healthy older adults Stage 1
Behavioral: Subtracting Cues training
  Arms: SCT healthy older adults Stage 2

SUMMARY:
Memory deficits are common after traumatic brain injuries (TBI) and are characteristic of various forms of dementia, such as Alzheimer's disease and its common precursor mild cognitive impairment (MCI). This project intends to assess the efficacy of cognitive rehabilitation in these patient populations. We will also use neuroimaging (functional magnetic resonance imaging - fMRI) to assess changes in brain activity that occur following cognitive rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria (all patients):

* A minimum of 12 years of education or attainment of a Graduation Equivalency Diploma;
* All medications stable for approximately 3 months;
* No history of severe mental illness;
* No current untreated alcohol or substance abuse/dependence;
* English as native and preferred language;
* MRI-compatible if taking part in fMRI studies 7) Able to give informed consent.

MCI Inclusion Criteria:

* Diagnosis of amnestic MCI based on criteria set forth by Petersen (2004). Additionally, other potential causes of cognitive deficit ruled out by the referring physician;
* 55 years of age or older.

TBI Inclusion criteria:

* History of a mild to moderate TBI;
* No history of other neurological disease or injury;
* A minimum of 6 months and maximum of 5 years post-onset of TBI;
* 18 - 45 years old.

Exclusion Criteria:

* History of neurological disease or injury (other than TBI)
* History of severe mental illness
* Current untreated alcohol or substance abuse
* Other conditions may exclude; please discuss with contact

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M. Hampstead, PhD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia, United States

REFERENCES:
- [Result] Hampstead BM, Sathian K, Phillips PA, Amaraneni A, Delaune WR, Stringer AY. Mnemonic strategy training improves memory for object location associations in both healthy elderly and patients with amnestic mild cognitive impairment: a randomized, single-blind study. Neuropsychology. 2012 May;26(3):385-99. doi: 10.1037/a0027545. Epub 2012 Mar 12. PMID 22409311

RESULTS

PARTICIPANT FLOW:
Groups:
- MST Healthy Older Adults: Stage 1: Mnemonic strategy training for object location associations for healthy older adults
- MST MCI: Stage 1: Mnemonic strategy training for object location associations in patients with MCI
- XP Healthy Older Adults: Stage 1: Repeated exposure for object location associations in healthy older adults
- XP MCI: Stage 1: Repeated exposure for object location associations in patients with MCI
- MST Healthy Older Adults: Stage 2: Mnemonic strategy training for face name associations in healthy older adults
- SCT Healthy Older Adults: Stage 2: Subtracting cues training for face name associations in healthy older adults
Period: Stage 1
Arm/Group | MST Healthy Older Adults: Stage 1 | MST MCI: Stage 1 | XP Healthy Older Adults: Stage 1 | XP MCI: Stage 1 | MST Healthy Older Adults: Stage 2 | SCT Healthy Older Adults: Stage 2
Started | 12 | 15 (11 allocated to intervention, but 1 withdrew before the first intervention session) | 11 | 14 | 0 | 0
Completed | 12 (1 patient excluded who completed training but did not disclose ongoing chemotherapy for cancer) | 15 | 10 | 14 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Period: Stage 2
Arm/Group | MST Healthy Older Adults: Stage 1 | MST MCI: Stage 1 | XP Healthy Older Adults: Stage 1 | XP MCI: Stage 1 | MST Healthy Older Adults: Stage 2 | SCT Healthy Older Adults: Stage 2
Started | 0 | 0 | 0 | 0 | 15 | 15
Completed | 0 | 0 | 0 | 0 | 15 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One participant from MST Healthy older adults Stage 1 excluded after study completion due to ongoing chemotherapy treatment (undisclosed during study).
  One participant from MST MCI Stage 1 excluded due to being diagnosed with Alzheimer's dementia within 1 month of completing study
Groups:
- Total: Total of all reporting groups
Arm/Group | MST Healthy Older Adults: Stage 1 | MST MCI: Stage 1 | XP Healthy Older Adults: Stage 1 | XP MCI: Stage 1 | MST Healthy Older Adults: Stage 2 | SCT Healthy Older Adults: Stage 2 | Total
Number analyzed (Participants) | 11 | 14 | 10 | 14 | 15 | 15 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (7.7) | 73.5 (10.1) | 72.5 (6.8) | 70.5 (5.8) | 67.1 (7.9) | 72.0 (7.6) | 71.3 (7.9)
Gender [Count of Participants; unit: Participants]
  Female | 7 | 4 | 6 | 8 | 13 | 13 | 51
  Male | 4 | 10 | 4 | 6 | 2 | 2 | 28
Region of Enrollment [Number; unit: participants]
  United States | 11 | 14 | 10 | 14 | 15 | 15 | 79

OUTCOME MEASURES:

1. Primary Outcome: Memory Test Accuracy on Trained Stimuli
Description: Accuracy (Percent correct) for trained stimuli. Stage 1: Object location association test Stage 2: Face name association test
Time Frame: Pre-training, post-training, 1 month
Population: MST older adults Stage 1: 1 participant excluded due to undisclosed ongoing chemotherapy treatment XP older adults Stage 1: 1 participant decided not to participate after randomization MST MCI Stage 1: 1 participant diagnosed with Alzheimer's dementia within 1 month of completing study
Measure: Mean (Standard Deviation); unit: Percent correct
Arm/Group | MST Healthy Older Adults: Stage 1 | MST MCI: Stage 1 | XP Healthy Older Adults: Stage 1 | XP MCI: Stage 1 | MST Healthy Older Adults: Stage 2 | SCT Healthy Older Adults: Stage 2
Number analyzed (Participants) | 11 | 14 | 10 | 14 | 15 | 15
Percent correct
  Pre-training | 53.9 (10.2) | 37.6 (15.0) | 48.9 (14.5) | 37.3 (8.7) | 59.8 (14.0) | 57.6 (15.3)
  Post-Training | 97.0 (4.0) | 82.5 (14.7) | 92.0 (6.9) | 71.4 (13.2) | 94.9 (4.8) | 83.7 (13.7)
  1-month: number analyzed (Participants) | 11 | 13 | 10 | 11 | 15 | 15
  1-month | 85.3 (1.01) | 65.1 (17.8) | 63.3 (13.7) | 45.8 (8.3) | 86.2 (7.4) | 69.7 (18.1)

ADVERSE EVENTS:
Arm/Group | MST Healthy Older Adults: Stage 1 | MST MCI: Stage 1 | XP Healthy Older Adults: Stage 1 | XP MCI: Stage 1 | MST Healthy Older Adults: Stage 2 | SCT Healthy Older Adults: Stage 2
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15 | 0/11 | 0/14 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/15 | 0/11 | 0/14 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes